CLINICAL TRIAL: NCT05250219
Title: Identifying and Quantifying Microchimeric Maternal Cells in Young Males, Potentially Acquired Through Breastfeeding - A Pilot Study
Brief Title: Microchimeric Cell Tranfer From Mother to Child - Pilo Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0724
Record Dates: First submitted 2018-12-24; First posted 2022-02-22 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2022-02

CONDITIONS: Breastfeeding
Keywords: Microchimeric; Microchimerism
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients for tonsils: 40 patients for tonsils
- patients for appendixes: 40 patients for appendixes)

SUMMARY:
Microchimeric cells are known to be transferred from mother to child through the placenta. However it has been postulated that they could also be transferred through breastfeeding.

This study is designed to analyse lymphoid and digestive tract tissues (tonsils and appendixes) in male infants (or young adults) to research microchimeric female cells and try to correlate the frequency and localisation of said cells to the breastfeeding status during early infancy

ELIGIBILITY:
Inclusion criteria:

* age 1-16 years (at the time of surgery)
* male
* known breastfeeding status in infancy

Exclusion criteria:

* premature birth (before 37 weeks)
* history of blood transfusion
* history of bone marrow transplant
* history of organ transplant
* patient known to have a twin
* known gonosomal

Ages: 1 Year to 16 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Study Population: Young males, undergoing surgery (appendectomy ou tonsillectomy) for medical reasons
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
To identify microchimeric cells of maternal origin in lymphoid | day 1
  To identify microchimeric cells of maternal origin in lymphoid in young males cytogenetic FISH staining, coupled with MS-PCR, to identify microchimeric cells.
To identify microchimeric cells of maternal origin in digestive tissues | day 1
  To identify microchimeric cells of maternal origin in digestive tissues in young males cytogenetic FISH staining, coupled with MS-PCR, to identify microchimeric cells.
to determine Quantifying the microchimeric cells | day 1
  Quantifying the microchimeric cells : Cell quantification will be assessed through FISH staining (automated cell counting) and qPCR
to determine locating the cells in tissues | day 1
  locating the cells in tissues : Appendix histology slides will be analysed after FISH staining to locate the microchimeric cells
to determine trying to find a correlation between breastfeeding status | day 1
  trying to find a correlation between breastfeeding status : Microchimeric cell quantification will be confronted to the breastfeeding status in infancy (collected during patient inclusion) to validate a correlation

CONTACTS AND LOCATIONS:
Overall Officials: Boris DMITRENKO, Study Director — UH MONTPELLIER - FRANCE
Locations (1):
- Uh Montpellier, Montpellier, France